CLINICAL TRIAL: NCT00155454
Title: Intravitreal Long Acting Gas in the Prevention of Early Postoperative Vitreous Hemorrhage in Diabetic Vitrectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 9461700621
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2012-12-27 (Estimated); Status verified 2012-12

CONDITIONS: Diabetes Mellitus; Diabetic Retinopathy; Vitreous Hemorrhage
Keywords: Diabetic retinopathy; Vitrectomy; Postoperative vitreous hemorrahge; Intravitreal gas injection
MeSH Terms: conditions — Diabetes Mellitus; Diabetic Retinopathy; Vitreous Hemorrhage

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Study group (Experimental): Group 1 had intravitreal long acting gas (10% C3F8) injection in the vitreous cavity at the end of surgery
  Interventions: Procedure: Intravitreal long acting gas (10% C3F8)
- Control group (Sham Comparator): Group 2 did not receive intravitreal long acting gas (10% C3F8)
  Interventions: Procedure: Intravitreal long acting gas (10% C3F8)

INTERVENTIONS:
Procedure: Intravitreal long acting gas (10% C3F8) — At the end of surgery, fluid-gas exchange with 10% C3F8 were done in the eye of study group

SUMMARY:
Recurrent vitreous hemorrhage after vitrectomy for complications of diabetic retinopathy is a common occurrence. The hemorrhage may appear within the first few weeks after surgery or months later. This complication may delay visual rehabilitation significantly and sometimes requires additional procedures or surgery, jeopardizing previous successful operation. The causes of bleeding are diverse. While evidence suggests fibrovascular proliferation from the sclerotomy sites or in the vitreous base may be an important source of recurrent vitreous hemorrhage, other origins of hemorrhage exist including lysed clot from residual vitreous skirt, injured retinal vessels from surgery, and incompletely removed fibrovascular tissues. The latter three conditions may be the major sources of early postoperative vitreous hemorrhage. We have shown that peripheral retinal cryotherapy along with cryo treatment at the sclerotomy sites may effectively reduce the incidence of fibrovascular proliferation at the inner surface of sclerotomy sites and prevent the late-onset recurrent vitreous hemorrhage. However, many patients still experience disturbing vitreous hemorrhage within the first two to three weeks after post-operative transient clear-up of the vitreous. We hypothesize that gas bubble within the vitreous cavity may mechanically temponade the fragile retinal vessels, and concentrate the coagulation factors in the vitreous cavity, allowing the integrity of vessel walls gradually recovers and thus preventing the occurrence of early postoperative recurrent vitreous hemorrhage.

To test this hypothesis, a clinical study was undertaken to investigate the effect of long-acting gas infused into the vitreous cavity at the end of diabetic vitrectomy in the prevention of recurrent vitreous hemorrhage.

DETAILED DESCRIPTION:
The study consisted of two parts. Part one was prospective clinical observational study; part two was case control study.

From January 2005 to May 2005, consecutive patients undergoing primary pars plana vitrectomy for complications of proliferative diabetic retinopathy were recruited for the prospective study. The selection criteria were: 1) anticoagulant therapy should not have been used prior to surgery or during post-operative follow-up period; 2) ther should be no medical history of blood diseases associated with abnormal blood coagulation. During operation, removal of the fibrovascular tissues as well as old and fresh blood was attempted as completely as could be safely done in all cases; blood clots adherent to the peripheral vitreous skirt was removed as much as possible; peripheral retinal cryotherapy (10 to 12 spots in one row), and sclerotomy sites cryo (2 spots, each 6 seconds, for 3 sclerotomy sites) were performed. For those cases without retinal detachment and breaks, fluid-gas exchange with 7.5% C3F8 was done at the end of the surgery; For those with preexisting breaks or iatrogenic breaks induced retinal detachment, fluid-gas exchange with 15% C3F8 was performed before cryotherapy. After surgery, patients without breaks were kept in a prone position overnight, and maintained head down during waking hours and lied on either side, during sleep for 3 weeks. Other patients assumed head positions depending on the location of breaks. Ophthalmological examinations were performed in the first 4 days after surgery, then weekly for 6 weeks and then monthly for 4 months. The preoperative, intraoperative and postoperative data were collected for each patient. These included age, gender, study eye, types and duration of diabetes mellitus, intraoperative diagnosis, and the use of scleral buckle, silicone oil temponade; data regarding the time, duration, frequency and treatment of recurrent vitreous hemorrhage and the duration of post-operation follow-up were also compiled. Results of ophthalmological examinations, including best corrected visual acuity, intraocular pressures, corneal conditions, anterior chamber reactions, lens status, intravitreal gas amount, and retina conditions were recorded. The amount of vitreous blood was assessed by indirect ophthalmoscopy with patients in both sitting and face-up position. The degree of vitreous opacity was recorded according to criteria set for grading vitreous opacity in uveitis.

Patients who had silicone oil infusion, failed to achieve retinal attachment for at least 3 months, or followed for less than a minimum of 5-month were excluded from the study.

Using the same inclusion and exclusion criteria, chart review from September 2004 to May 2005 for diabetic cases operated by the same surgeon with only cryo treatment but without long-acting gas infusion at the end of vitrectomy was done. Similar data as for the prospective study (except intravitreal gas amount) were collected. These cases served as control to compare the rate of recurrent vitreous hemorrhage and the change of best-corrected visual acuity between cases with intravitreal long-acting gas and those without.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing primary pars plana vitrectomy for complications of proliferative diabetic retinopathy were recruited for the prospective study

Exclusion Criteria:

* (1) anticoagulant therapy had been used prior to surgery or during post-operative follow-up period; (2) positive medical history of blood diseases associated with abnormal blood coagulation.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2004-09; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Recurrent vitreous hemorrhage rate | Within 6 months after vitrectomy
  Initial time to vitreous clearing , percentage of prolonged vitreous clearing, and early versus late manifest postoperative recurrent vitreous hemorrhage in groups 1 and 2 were compared to determine the effects of long acting gas on prevention of early recurrent vitreous hemorrhage.

CONTACTS AND LOCATIONS:
Overall Officials: Chung-May Yang, MD, Study Director — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan